CLINICAL TRIAL: NCT05382013
Title: Efficacy and Safety of Avatrombopag for Treating Thrombocytopenia in Hepatitis b Virus Related Acute-on-chronic Liver Failure Patients Receiving Artificial Liver Support System Treatment
Brief Title: Efficacy and Safety of Avatrombopag for Treating TCP in HBV-ACLF Patients Receiving ALSS Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PL16
Record Dates: First submitted 2022-05-14; First posted 2022-05-19 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Thrombocytopenia; Hepatitis B, Chronic; Acute-On-Chronic Liver Failure
Keywords: thrombocytopenia; hepatitis B virus; acute-on-chronic liver failure; double plasma molecular adsorption system; plasma exchange; artificial liver support system
MeSH Terms: conditions — Thrombocytopenia; Hepatitis B, Chronic; Acute-On-Chronic Liver Failure; Hepatitis B | interventions — avatrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trial Group (Experimental): 30 patients receive treatment of avatrombopag, DPMAS, LPE, and comprehensive internal medical treatment.
  Interventions: Drug: Avatrombopag; Other: Artificial Liver Support System; Other: Comprehensive internal medical treatment.
- Control Group (Active Comparator): 30 patients receive treatment of DPMAS, LPE, and comprehensive internal medical treatment.
  Interventions: Other: Artificial Liver Support System; Other: Comprehensive internal medical treatment.

INTERVENTIONS:
Drug: Avatrombopag — Patients will receive treatment of oral avatrombopag 20mg per day for the first 5 days
  Arms: Trial Group
Other: Artificial Liver Support System — Patients will receive treatment of double plasma molecular adsorption system (DPMAS) and low volume plasma exchange (LPE) for three times. The volume of plasma adsorption in DPMAS is 5000~6000 millilitre. The volume of fresh frozen plasma used in LPE is 1000 millilitre.
Other: Comprehensive internal medical treatment. — Patients will receive comprehensive internal medical treatment.

SUMMARY:
This study aims to investigate the efficacy and safety of avatrombopag for treating thrombocytopenia in hepatitis b virus related acute-on-chronic liver failure patients receiving artificial liver support system treatment.

DETAILED DESCRIPTION:
Artificial liver support system (ALSS) is an optimal therapy in patients with hepatitis b virus (HBV) related acute-on-chronic liver failure (ACLF). But a lot of patients encount thrombocytopenia (TCP) due to the mechanical damage of thrombocyte and use of heparin during the treatment. Avatrombopag is an oral thrombopoietin receptor agonist that has been recently approved for treating TCP in chronic liver disease patients needing invasive procedures. Therefore, this study aims to investigate the efficacy and safety of avatrombopag for treating TCP in HBV related ACLF patients receiving ALSS treatment. Sixty patients with HBV related ACLF receiving ALSS will be enrolled in this study. The participants are divided into trial group (avatrombopag, double plasma molecular adsorption system (DPMAS) , low volume plasma exchange (LPE), and comprehensive internal medical treatment) and control group (DPMAS, LPE, comprehensive internal medical treatment). Symptoms, signs, laboratory tests results, adverse events, mortality rates are recorded from treatment baseline to 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65 years old;
2. Clinical diagnosis of chronic hepatitis b virus infection (positive hepatitis b surface antigen or positive hepatitis b virus DNA > 0.5 year);
3. Clinical diagnosis of liver failure (serum total bilirubin level > 10 times upper limit of normal; prothrombin time activity < 40% and ≥20%, or prothrombin time international ratio ≤ 2.6 and > 1.5);
4. Platelets < 80*10 E9/L and > 50*10 E9/L.
5. Signed informed consent form.

Exclusion Criteria:

1. Other active liver diseases;
2. Hepatocellular carcinoma or other malignancy;
3. Pregnancy or lactation;
4. Human immunodeficiency virus infection or congenital immune deficiency diseases;
5. Severe diabetes, autoimmune diseases; unstable infarction due to cardio-cerebrovascular events; other important organ dysfunctions or transplantation;
6. Severe complications including severe infection, gastrointestinal bleeding, hepatic encephalopathy, hepatorenal syndrome;
7. Patients with ALSS treatment in one week;
8. Thrombotic disease;
9. Patients can not follow-up;
10. Investigator considering inappropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of platelet ≥50*10E9/L | 3 weeks
  Rate of patients with platelet ≥50*10E9/L during ALSS treatment

SECONDARY OUTCOMES:
Rate of bleeding | 3 weeks
  Incident rate of patients with bleeding during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, results and conclusions of this clinical trial will be published at academic conferences or in journals.
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to pliang@mail.sysu.edu.cn. To gain access, data requestors will need to sign a data access agreement.